CLINICAL TRIAL: NCT05905081
Title: Acute Effects of Physical Fitness and Aerobic Exercise on Cognitive Functions in Young Adult Males
Brief Title: Acute Effects of Moderate Intensity Aerobic Exercise on Cognitive Functions in Young Adult Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Şermin Tükel Akay, Asst. Prof., Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 4930-GOA
Record Dates: First submitted 2023-05-03; First posted 2023-06-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Change
Keywords: acute aerobic exercise; cognition; university students; physical fitness
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two group comparison, before and after intervention
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): 30-minutes moderate-intensity aerobic exercise will be performed according to ACSM guidelines
  Interventions: Other: aerobic exercise
- Control Group (No Intervention): 30-minutes video screening while sitting

INTERVENTIONS:
Other: aerobic exercise — 30-minutes aerobic exercise intervention on the bicycle ergometer. The exercise protocol includes 5 minutes of warm-up, 20 minutes of loading and 5 minutes of cool-down. The intensity of the exercise will be adjusted to be between 46% and 63% of the VO2max calculated according to the exercise programming guide published by the American College of Sports Medicine (ACSM), and the perceived effort level on the Borg scale will be 12-13. Warm-up and cool-down periods will be set to 46% of VO2max and Borg perceived exertion level below 9.
  Arms: Exercise Group

SUMMARY:
60 healthy male university students will be included in this study. Physical fitness parameters, fluid intelligence, and physical activity level will be measured at baseline. Participants will be randomised to one of two testing schedules, groups will complete either a 30-minutes aerobic exercise session or a resting control condition. Cognitive measures (simple reaction time task, go/nogo task, spatial cueing, n-back task) will be tested before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* No known psychiatric, cognitive or physical health problems
* No limiting issue for performing exercise according to Physical Activity Readiness Questionnaire (PAR-Q+)
* Physical activity level according to International Physical Activity Questionnaire (IPAQ) < 3000 MET

Exclusion Criteria:

* Discomfort/illness that will interfere with physical activity
* Using any medication or stimulants
* Having limitations for performing exercise according to Physical Activity Readiness Questionnaire (PAR-Q+)

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in motor inhibition | Baseline and 30 mins after baseline
  Go/NoGo Task
Change in working memory capacity | Baseline and 30 mins after baseline
  N-Back Task

SECONDARY OUTCOMES:
Change in psychomotor rate | Baseline and 30 mins after baseline
  Simple reaction time task
Change in visual inspection and attention | Baseline and 30 mins after baseline
  Spatial cueing

OTHER OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | At baseline
  IPAQ score under 300 indicates low physical activity, 300-3000 indicates moderate physical activity and higher than 3000 is high physical activity.
VO2max | At baseline
  Astrand test
Raven's Progressive Matrices | At baseline
  Fluid intelligence
Muscle strength | At baseline
  back-chest-leg strength
Plank test | At baseline
  muscular endurance
T-test | At baseline
  agility
Body composition | At baseline
  Body Mass Index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Şermin Tükel Akay, PhD, Principal Investigator — Izmir University of Economics
Locations (1):
- Izmir University of Economics, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No